CLINICAL TRIAL: NCT03377153
Title: Evaluation of the Effects of Hesperidin and Flaxseed Supplementation on Hepatic Enzymes, Inflammatory Factors, Lipid Profile, Blood Glucose, Insulin Sensitivity, and Hepatic Steatosis Grade in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: The Effects of Hesperidin and Flaxseed on Biochemical Factors and Hepatic Fibrosis in Nonalcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6757
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-04

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Hesperidin; Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hesperidin and Flaxseed (Active Comparator)
  Interventions: Dietary Supplement: hesperidin and flaxseed
- control (Placebo Comparator)
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: hesperidin and flaxseed — 2 capsuls hesperidin and 30 g flaxseed
  Arms: Hesperidin and Flaxseed
Other: control — no supplementation
  Arms: control

SUMMARY:
To study the effects of Hesperidin and flaxseed supplement on lipid profile, liver enzymes, inflammatory factors and hepatic fibrosis in patients with Nonalcoholic Steatohepatitis (NASH), 50 patients who referred to Gastrointestinal (GI) clinic with steatosis grade 2 and 3 will be randomly allocated to contol group or 2 capsules Hesperidin and 30 gram flaxseed for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, lipid profiles, liver enzymes, some inflammatory markers, and liver fibrosis will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

- Age of 18 to 70 years

* Body Mass Index (BMI) between 25-40
* Sonographic findings compatible with hepatic steatosis (degree 2 or more)

Exclusion Criteria:

* Diabetes
* Taking any kind of antibiotics two weeks before recruitment
* History of alcohol consumption
* pregnancy or lactation
* Professional athletes
* Other liver disease (viral/etc)
* Use of drugs such as calcium channel blockers, high dose synthetic estrogens, methotrexate , amiodarone, steroids, chloroquine, immunosuppressive drugs, lipid-lowering agents, metformin and vitamin E
* A history of Hypertension, Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* History of Upper GI surgery / Prior surgical procedures such as jejunoileal or jejunocolic bypass, gastroplasty
* Following program to lose weight in recent 3 mo
* A history of hypothyroidism or Cushing's syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
liver fibrosis | 12 weeks
  assess by fibroscan

SECONDARY OUTCOMES:
body mass index | 12 weeks
  is universally expressed in units of kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran